CLINICAL TRIAL: NCT02595749
Title: Effects of Intranasal Oxytocin on Cigarette Smoking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Matthew Kirkpatrick, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-15-00657
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Nicotine Dependence; Tobacco Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo then Intranasal Oxytocin (40 IU) (Experimental): Participants received a single placebo nasal spray (consisting of 4ml sterile saline [Ocean Nasal Spray Solution]) during the first experimental session, which occurred on a single day. After a 72 hour washout period, they then received a single 40 IU dose of Pitocin (oxytocin, USP; concentration = 10 IU/1 mL; PAR Pharmaceuticals, NY, USA) during the second experimental session, which occurred on a single day. All nasal spray solutions were transferred into two, 2 ml intranasal atomizers and administered in four sprays to each nostril over the course of 10 minutes.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Intranasal Oxytocin (40 IU) then Placebo (Experimental): Participants received a single 40 IU dose of Pitocin (oxytocin, USP; concentration = 10 IU/1 mL; PAR Pharmaceuticals, NY, USA) during the first experimental session, which occurred on a single day. After a 72 hour washout period, they then received a single placebo nasal spray (consisting of 4ml sterile saline [Ocean Nasal Spray Solution]) during the second experimental session, which occurred on a single day. All nasal spray solutions were transferred into two, 2 ml intranasal atomizers and administered in four sprays to each nostril over the course of 10 minutes.
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Pitocin
Drug: Placebo
  Other Names: Ocean Spray saline spray

SUMMARY:
Socioemotional processing dysfunctions (i.e., disruptions in affective, cognitive, and neural processes that encode, interpret, and respond to socially and emotionally relevant stimuli) have been implicated in tobacco smoking and relapse, however this potential target for medication development has not been systematically examined. Evidence from animal and human laboratories indicate that administration of intranasal oxytocin enhances socioemotional processing and may be efficacious for the treatment of drug addiction, including nicotine dependence. In order to evaluate the potential efficacy of intranasal oxytocin for smoking cessation, this laboratory-based proposal will examine whether intranasal oxytocin attenuates smoking lapse, nicotine withdrawal, and socioemotional processing disruptions in regular smokers following overnight abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-40
* Smoke >= 10 cig/day for the past year
* English fluency

Exclusion Criteria:

* Current DSM-5 substance use disorder, excluding nicotine dependence (to minimize alcohol or drug withdrawal symptoms during the study sessions)
* Any medical condition that would increase risk for study participation (such as sinus infection or other condition blocking access to the olfactory epithelium)
* Women who are pregnant or nursing
* Current use of psychiatric medication
* Breath Carbon Monoxide (CO) levels < 10ppm measured during study intake (to exclude individuals who overreport smoking in order to participate in the study)
* Planning to quit or reduce smoking in the next 30 days
* Current regular use of other nicotine products

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kirkpatrick, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC Health, Emotion and Addiction Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were excluded pre-assignment.
Groups:
- Placebo Then Intranasal Oxytocin (40 IU): Participants received a single placebo nasal spray (consisting of 4ml sterile saline [Ocean Nasal Spray Solution]) during the first experimental session, which occurred on a single day. After a 72 hour washout period, they then received a single 40 IU dose of Pitocin (oxytocin, USP; concentration = 10 IU/1 mL; PAR Pharmaceuticals, NY, USA) during the second experimental session, which occurred on a single day. All nasal spray solutions were transferred into two, 2 ml intranasal atomizers and administered in four sprays to each nostril over the course of 10 minutes.
  Oxytocin
Period: Overall Study
Arm/Group | Placebo Then Intranasal Oxytocin (40 IU) | Intranasal Oxytocin (40 IU) Then Placebo
Started | 45 | 38
Completed | 33 | 31
Not Completed | 12 | 7
Not completed — Withdrawal by Subject | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Intranasal Oxytocin (40 IU) | Intranasal Oxytocin (40 IU) Then Placebo | Total
Number analyzed (Participants) | 45 | 38 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (5.4) | 29.8 (5.4) | 30.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 10 | 13
  Not Hispanic or Latino | 42 | 28 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 18 | 37
  White | 13 | 9 | 22
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 45 | 38 | 83

OUTCOME MEASURES:

1. Primary Outcome: Smoking Lapse Analogue Task (Delay Score)
Description: This task measures ability to resist the temptation to initiate smoking under conditions in which it is advantageous to remain abstinent. The "delay score" is the number of minutes before participants begin smoking (minimum = 0 minutes to maximum = 50 minutes). A higher number is better.
Time Frame: 2.5 hours after nasal spray administration
Measure: Mean (Standard Error); unit: minutes
Groups:
- Intranasal Oxytocin (40 IU): Participants received a single 40 IU dose of Pitocin (oxytocin, USP; concentration = 10 IU/1 mL; PAR Pharmaceuticals, NY, USA) during the first or second experimental session. The second experimental session was completed at least 72 hours after the first. All nasal spray solutions were transferred into two, 2 ml intranasal atomizers and administered in four sprays to each nostril over the course of 10 minutes.
- Placebo: Participants received a single placebo nasal spray (consisting of 4ml sterile saline [Ocean Nasal Spray Solution]) during the first or second experimental session. The second experimental session was completed at least 72 hours after the first. All nasal spray solutions were transferred into two, 2 ml intranasal atomizers and administered in four sprays to each nostril over the course of 10 minutes.
Arm/Group | Intranasal Oxytocin (40 IU) | Placebo
Number analyzed (Participants) | 64 | 64
minutes | 11.5 (2.3) | 10.9 (2.3)

2. Primary Outcome: Brief Questionnaire of Smoking Urges (QSU)
Description: The Brief Questionnaire of Smoking Urges (QSU) is a 10-item self-report questionnaire measures desire, intention, urge, and need to smoke. The QSU was assessed 30 minutes before the nasal spray, and again 30, 60, and 90 minutes after the nasal spray during each session. Scores at each assessment time are calculated as the mean of all 10 items (minimum = 0 to maximum = 5). Each session's scores are then calculated as the mean scores of post-spray assessments. A lower score is better.
Time Frame: 30 minutes before nasal spray, and 30, 60, and 90 minutes after nasal spray
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Oxytocin (40 IU) | Placebo
Number analyzed (Participants) | 64 | 64
score on a scale | 2.46 (0.12) | 2.49 (.11)

3. Primary Outcome: Systolic Blood Pressure (mmHg)
Description: Systolic blood pressure (SP) was assessed 30 minutes before the nasal spray, and again 30, 60, and 90 minutes after the nasal spray during each session. Each session's values are calculated as the mean of post-spray assessments.
Time Frame: 30 minutes before nasal spray, and 30, 60, and 90 minutes after nasal spray
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Intranasal Oxytocin (40 IU) | Placebo
Number analyzed (Participants) | 64 | 64
mmHg | 122.1 (1.4) | 118.2 (1.4)

4. Primary Outcome: Diastolic Blood Pressure (mmHg)
Description: Diastolic blood pressure (DP) was assessed 30 minutes before the nasal spray, and again 30, 60, and 90 minutes after the nasal spray during each session. Each session's values are calculated as the mean of post-spray assessments.
Time Frame: 30 minutes before nasal spray, and 30, 60, and 90 minutes after nasal spray
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Intranasal Oxytocin (40 IU) | Placebo
Number analyzed (Participants) | 64 | 64
mmHg | 77.5 (1.1) | 74.7 (1.1)

5. Primary Outcome: Heart Rate (Bpm)
Description: Heart rate (HR) was assessed 30 minutes before the nasal spray, and again 30, 60, and 90 minutes after the nasal spray during each session. Each session's values are calculated as the mean of post-spray assessments.
Time Frame: 30 minutes before nasal spray, and 30, 60, and 90 minutes after nasal spray
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Intranasal Oxytocin (40 IU) | Placebo
Number analyzed (Participants) | 64 | 64
bpm | 65.6 (0.7) | 65.9 (0.7)

6. Secondary Outcome: Profile of Mood States (Anxious Scale)
Description: The Profile of Mood States (POMS) lists 72 affective adjectives that are rated on 0 to 4-point. The main measure for this study is the Anxious scale, calculated as the mean of 6 anxiety-related items. The POMS was assessed 30 minutes before the nasal spray, and again 30, 60, and 90 minutes after the nasal spray during each session. Each session's scores are calculated as the mean scores of post-spray assessments. Lower scores are better.
Time Frame: 30 minutes before nasal spray, and 30, 60, and 90 minutes after nasal spray
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Oxytocin (40 IU) | Placebo
Number analyzed (Participants) | 64 | 64
score on a scale | 0.82 (.04) | 0.71 (.04)

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information in the current study did not differ from the clinicaltrials.gov definitions. Participants were monitored during experimental sessions in person and then for a week following study participation (by phone call each day).
Arm/Group | Intranasal Oxytocin (40 IU) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT02595749/Prot_SAP_000.pdf